CLINICAL TRIAL: NCT03757728
Title: Hemorrhoidal Pedicle Ligation vs Laser Hemorrhoidectomy vs Open Hemorrhoidectomy: Randomized, Double Blind, Multicenter Trial
Brief Title: Randomized Trial :Hemorrhoidal Pedicle Ligation vs Laser vs Open Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vilnius University (Other)
Collaborators: Biolitec Pharma Ltd. (Industry)
Responsible Party: Principal Investigator, Tomas Poskus, Professor, Vilnius University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 158200-15-792-322
Record Dates: First submitted 2018-11-18; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Hemorrhoids Second Degree; Hemorrhoids Third Degree

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- open haemorrhoidectomy (Other): Open haemorrhoidectomy is performed using an anal retractor, exposed haemorrhoids at 3 - 7- 11 hours are excised using cautery. The arteries are ligated or cauterized. Open or closed technique is used (the choice of the surgeon). The Spongostan plug is then introduced
  Interventions: Procedure: Haemorrhoidectomy operations
- Haemorrhodal pedicle ligation (Other): Haemorrhodal pedicle ligation is performed using operating proctoscope. The pedicle of symptomatic haemorrhoid is suture ligated with absorbable Vycril 2/0. Mucopexy is performed simultaneously if the prolapse is noticed. No tissue removal is performed
  Interventions: Procedure: Haemorrhoidectomy operations
- Intrahaemoroidal laser coagulation (Other): Intrahaemoroidal laser coagulation is performed using disposable THD kit [Biolitec Co]. The haemorrhoidal pedicle is sutured. 1mm opening is created at the external haemorrhoid (skin level). Laser is then introduced up to pedicle and coagulation performed. This is repeated to all the piles. The procedure is finished with placing Spongostan plug into anal canal
  Interventions: Procedure: Haemorrhoidectomy operations

INTERVENTIONS:
Procedure: Haemorrhoidectomy operations — for treatment of symptomatic 2 to 3 degree haemorrhoids

SUMMARY:
The aim of this study is to compare three different modalities for treatment of symptomatic 2 ° to 3 ° haemorrhoids: open haemorrhoidectomy, intrahaemorrhoidal laser procedure and haemorrhoidal pedicle ligation.

To assess early outcomes (after one week and one month) of the procedures: pain, bleeding, wound healing, return to work and quality of life; To assess late outcomes (after one year) of the procedures: late functional results (continence) and recurrence of symptoms and haemorrhoids.

Study design This is a multi-center, double-blind, prospective RCT comparing three different modalities for treatment of symptomatic 2 ° to 3 ° haemorrhoids: open haemorrhoidectomy, intrahaemorrhoidal laser coagulation and haemorrhoidal artery ligation.

DETAILED DESCRIPTION:
Hemorrhoidal pedicle ligation vs laser hemorrhoidectomy vs open hemorrhoidectomy: randomized, double blind, multicenter trial

AIMS AND OBJECTIVES The aim of this study is to compare three different modalities for treatment of symptomatic 2 to 3 ° haemorrhoids: open haemorrhoidectomy, intrahaemorrhoidal laser procedure and haemorrhoidal pedicle ligation.

Objectives of the study are:

To assess early outcomes (after one week and one month) of the procedures: pain, bleeding, wound healing, return to work and quality of life; To assess late outcomes (after one year) of the procedures: late functional results (continence) and recurrence of symptoms and haemorrhoids.

MATERIALS AND METHODS Study design This is a randomized, parallel group (1:1:1) double-blinded single centre prospective study. No changes in methods of the study were allowed after commen cement. This RCT compares three different modalities for treatment of symptomatic 2 to 3 ° haemorrhoids: open haemorrhoidectomy, intrahaemorrhoidal laser coagulation and haemorrhoidal artery ligation.

Patients This prospective randomized study was performed at Vilnius University Hospital Santara Clinics, Vilnius, Lithuania. It is a large tertiary University hospital with dedicated outpatient clinic. A period of 3 year starting from April 2015 to November 2018. A total of 121 patients are included in the study.

Patients with symptomatic 2nd or 3rd ° hemorrhoids, in 1st or 2nd risk group of ASA (American Society of Anesthesiologists), who consented to participate in this study were included into the study. Exclusion criteria were 1st or 4th °of hemorrhoids, pregnancy, patients with other anorectal diseases (fistula, abscess, rectal carcinoma, inflammatory bowel disease, etc.), patients after previous anal operations (except rubber band ligation, which should have occurred more than 3 months before the inclusion in the trial) and ≥ 3rd risk group of ASA.

Preoperative evaluation Detailed physical and anorectal examination was performed with anoscopy and rigid proctoscopy in all cases, as well as colonoscopy if indicated. All patients filled a dedicated symptom questionnaire, which included questions on intensity and frequency of hemorrhoidal prolapse, bleeding, itching, pain and other symptoms. Every patient completed Wexner incontinence score and SF-36 questionnaires.

Preoperative examination, classification, operation technique, postoperative treatment and follow-up are discussed at the introductory course.

Patients preoperatively fill questionnaires on the quality of life and defecation function (Patient symptoms scale, Cleveland clinic incontinence scale, Health survey - SF 36, Fecal incontinence quality of life instrument - FIQol).

Patient symptoms scale (appendix 1) - symptoms of haemorrhoids are assessed (rectal bleeding, pain, pile prolapse, defecation disturbances, discomfort affecting normal life). Each symptom gets a number from 1 - very intense to 5 - no complaints.

Cleveland clinic incontinence scale (appendix 2) - the sum of 5 parameters is determined that are scored on a scale from 0 (=absent) to 4 (daily) frequency of incontinence to gas, liquid, solid, of need to wear pad, and of lifestyle changes. A score of 0 means perfect control, a score of 20 - complete incontinence.

Health survey - SF 36 (appendix 3) - it measures eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health. For each of the eight domains that the SF36 measures an aggregate percentage score is produced. The percentage scores range from 0% (lowest or worst possible level of functioning) to 100% (highest or best possible level of functioning).

Fecal incontinence quality of life instrument - FIQol (appendix 4) -scale consists of 29 questions in 4 domains: lifestyle, coping/behavior, depression/self perception, embarrassment. Category ranges: 1 to 4 for lifestyle, coping/behavior, and embarrassment; 1 to 6 for depression/self perception.

Randomization, blinding and concealment The patients were randomized into three groups. Randomization sequence was computer-generated before the start of the trial. Every consecutive case

-history was assigned a randomization number (1, 2 or 3). It was written and sealed within the envelope and remained unknown neither to the patient, nor to the treating physician, to avoid selection bias. In the operating room, after induction of anesthesia, operating room junior staff was asked to unseal the envelope and the intervention was performed according to the procedure assigned. Pre- and postoperative patient management was identical in all three operations. The patient remained unaware of the procedure performed until the end of the study 1 year after the operation. The case-notes and discharge summary of the patient contained only the note, saying that the patient is included in the study of hemorrhoids with D.Danys/T.Poskus as Principal Investigators, patient's number is X. This number was within the locked and coded database and the staff, evaluating the result of the patients' treatment remained unaware of the procedure allocated. The patients were followed-up by different surgeons (E.P. and V.J.) than the ones, performing the operation. They had the access to the patient notes but not to the coded database, and were not able to know, which procedure was performed. In emergency situations, un-blinding of the patient and treating physicians was possible but was not required in any of the patients.

Operative procedure Patients were started on lactulose the day before the operation, which was continued after the operation to have regular bowel movements. Preoperative intravenous antibiotic prophylaxis was given according to the hospital protocol, which was 1g of Cephazolin (2g if patient was over 80 kg of weight), 240 mg of gentamycin and 500 mg of metronidazole (Ciprofloxacin can be used if patient is allergic to cephalosporins). Each surgeon performing operative procedures (T.P., D.D. and S.M.) had personal experience of at least 50 operations of each modality. 1 hour seminar was conducted between all surgeons before the start of the trial to unify the technique of operative procedures.All patients were photographed after induction of anesthesia before the start of the procedure and immediately after the procedure.LHP was performed using Ceralas diode laser of 1420 nm wavelength (Biolitec). Disposable LHP kit (Biolitec) was used, which contains sharp-tipped laser fiber and anoscope. Perianal skin immediately aboral to hemorrhoid was penetrated using needle-tip cautery (Figure 2). Laser fiber was introduced into the opening until the level of hemorrhoidal pedicle and coagulation was activated. 8 Watt 3 second pulses with 1 second pulse-pauses were used to coagulate the area of hemorrhoids. 5 mm of hemorrhoidal tissue is coagulated with one such pulse (experimental data). 250 Joules was the upper limit of energy delivered per 1 hemorrhoidal quadrant. Smaller hemorrhoids were treated with less energy, larger ones - with more energy. The procedure was repeated in three other quadrants, thus treating all anal circumference. RAR was performed as described by Schurmann JP et al. For these patients, the ligations were placed in the area of visible pathologic hemorrhoidal tissue, and in patients with large prolapse mucopexy - lifting of prolapsing hemorrhoidal tissue with sutures was performed. Standard EH was performed up to the level of hemorrhoidal pedicle, with ligation or suture-ligation of the pedicle and meticulous hemostasis. Follow-up was performed by different surgeons to those, performing the operations (E.P., V.J.). Each of them has more than 25 years of experience of colorectal and hemorrhoidal surgery. 1 hour seminar was conducted with them to unify the evaluation of the patients within the study. Each patient was followed up at 1 and 6 weeks and after 1 year after the operation (Figure 1). Perianal examination with photographic documentation was performed during all the visits. Anoscopy was performed during visits at 6 weeks and 1 year. Each patient was asked to fill in the diary during each day of the first post-operative week and present it at the first visit after 1 week. Symptom questionnaires were filled in during visits at 1 and 6 weeks and 1 year. Wexner incontinence score was filled during the visit at 6 weeks and 1 year. SF-36 QOL questionnaire was filled during the final visit at 1 year.

Statistical analysis Sample size calculation was performed using R statistical software package(©The R Foundation).Presuming the effect size of 0.3, power of 0.8 and alpha=0.05 the sample size was calculated to be 108 patients. To compensate for possible follow-up losses sample size was increased to 120 patients. Chi-square test and Anova tests were used to compare differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* All consented >18 year old male and female patients with 2 to 3 degree

Exclusion Criteria:

1. Patients with 1st and 4th degree haemorrhoids.
2. Patients with associated anorectal pathology (anorectal fistula, abscess, fissure, tumor or inflammatory bowel disease).
3. Patients who had undergone previous anorectal surgery.
4. ASA > 3.
5. Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of rectal prolapse | one years
  Visual rectal prolapse during postoperative anoscopy requiring any kind of medical attention or treatment (visit to the doctor or pharmacy, medical, invasive or surgical treatment).
Recurrence rate of rectal bleeding | one years
  Intensity and frequency of postoperative bleeding requiring any kind of medical attention or treatment (visit to the doctor or pharmacy, medical, invasive or surgical treatment).

SECONDARY OUTCOMES:
Continence | after one year
  Using Wexner fecal incontinence score (Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum 1993; 36:77-97)
Recurrence of any perianal symptoms | One years
  Evalluation by abdominal surgeon: pain, bleeding, external haemorrhoids, etc
Time to return to work | One years
  Time to return to work or regular activity, in days, reported by the patient
Intensity and duration of postoperative perianal pain | 7 postoperative days
  Intensity and duration of perianal pain after the operation (in days) based on visual analogue scale during after first 7 days of the operation
Quality of life | One years
  Quality of life based on Short-form (SF)-36 questionnaire (https://www.rand.org/health/surveys_tools/mos/36-item-short-form.html )
Fecal incontinence quality of life (FIQOL) score | One years
  Fecal incontinence quality of life (FIQOL) score at 1 year (Rockwood TH, Church JM, Fleshman JW. Fecal incontinence quality of life scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum 2000; 43:9-17)
Evaluation of the operation by the patient | One years
  Evaluation of the operation by the patient on visual analogue scale from 1 to 10 at 1-year visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Abdominal Surgery, Vilnius University Hospital Santariskiu Clinics, Lithuania, 2 Santariskiu Street,, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
2017